CLINICAL TRIAL: NCT06936566
Title: Phase 2 Study of Ruxolitinib-Based Primary Treatment for Acute GVHD
Brief Title: MAGIC Ruxolitinib for aGVHD
Acronym: MAGIC V
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: John Levine (Other)
Collaborators: Incyte Corporation (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, John Levine, Professor of Internal Medicine and Pediatrics, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-24-01656; P01CA039542 (NIH)
Record Dates: First submitted 2025-04-12; First posted 2025-04-20 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Acute Graft-versus-host Disease; Allogeneic Bone Marrow Transplantation; Adverse Effects
MeSH Terms: interventions — ruxolitinib; Methylprednisolone; Methylprednisolone Acetate; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Minnesota Standard Risk lower dose (Experimental): Patients receive lower dose ruxolitinib orally (PO) twice daily (BID) for 56 days then begin taper PO once daily (QD) for 1 week in the absence of disease progression or unacceptable toxicity
  Interventions: Drug: Ruxolitinib
- Minnesota Standard Risk higher dose (Experimental): Patients receive higher dose ruxolitinib PO BID for 56 days then begin taper PO BID for 1 week, followed by PO QD for 1 week in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ruxolitinib
- Minnesota High Risk (Experimental): Patients receive higher dose ruxolitinib PO BID for 56 days then begin taper PO BID for 1 week, followed by PO QD for 1 week in the absence of disease progression or unacceptable toxicity. Patients also receive systemic corticosteroid (methylprednisolone or similar) for a minimum of 3 days, then taper dose every 3-5 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ruxolitinib; Drug: Methylprednisolone

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib twice daily for 56 days followed by a short taper Given orally
  Other Names: Jakafi
Drug: Methylprednisolone — Starting dose 2 mg/kg/d for at least three days, then taper Given IV or orally
  Other Names: Depo-Medrol; Medrol; Solu-Medrol
  Arms: Minnesota High Risk

SUMMARY:
This clinical trial will study ruxolitinib-based treatment of acute graft-versus-host-disease (GVHD) that developed following allogeneic hematopoietic cell transplant. Acute GVHD occurs when donor cells attack the healthy tissue of the body. The most common symptoms are skin rash, jaundice, nausea, vomiting, and/or diarrhea. The standard treatment for GVHD is high dose steroids such as prednisone or methylprednisolone, which suppresses the donor cells, but sometimes there can be either no response or the response does not last. In these cases, the GVHD can become dangerous or even life threatening. High dose steroid treatment can also cause serious complications. Researchers have developed a system, called the Minnesota risk system, to help predict how well the GVHD will respond to steroids based on the symptoms present at the time of diagnosis. The Minnesota risk system classifies patients with newly diagnosed acute GVHD into two groups with highly different responses to standard steroid treatment and long-term outcomes. This protocol maximizes efficiency because all patients with grade II-IV GVHD are eligible for screening and treatment is assigned according to patient risk. Patients with lower risk GVHD, Minnesota standard risk, have high response rates to steroid treatment. In this trial the researchers will test whether ruxolitinib alone is as effective (non-inferior) as steroid-free therapy and safe. Patients will be randomized to two different doses of ruxolitinib to identify the dose which maximizes efficacy while minimizing toxicities such as hematologic and infectious toxicities. Patients with higher risk GVHD, Minnesota high risk, have unacceptable outcomes with systemic corticosteroid treatment alone and the researchers will test whether adding ruxolitinib, a proven effective second line GVHD treatment, can improve outcomes when added to systemic corticosteroids as first line treatment.

ELIGIBILITY:
Inclusion Criteria:

* Standard risk cohort: Minnesota standard risk GVHD (except patients with grade I [<50% BSA rash])
* High risk cohort: Minnesota high risk GVHD 3 GVHD that developed after DLI for mixed chimerism or poor graft function is allowed
* No prior systemic acute GVHD treatment. Topical or non-absorbed steroids are permitted.
* All donor types, HLA-matches, conditioning regimens, or GVHD prophylaxis strategies are acceptable
* ≥18 years of age
* Standard risk cohort: Hematopoietic engraftment with absolute neutrophil count (ANC) ≥ 1000/μL and platelet count ≥20,000. Use of growth factor supplementation and transfusions to maintain adequate hematologic parameters are allowed.
* High risk cohort: Hematopoietic engraftment with ANC ≥ 500/uL and platelet count ≥20,000. Use of growth factor supplementation and transfusions to maintain adequate hematologic parameters are allowed.

Exclusion Criteria:

* Systemic treatment with ruxolitinib or any other JAK inhibitor within 7 days of study entry
* Prior use of ruxolitinib to treat GVHD at any time
* Relapsed, progressing or persistent malignancy requiring withdrawal of systemic immunosuppression
* Relapse prior to development of GVHD unless subsequently in remission for at least 3 months
* GVHD that developed after DLI for relapse is not allowed without study PI or medical monitor approval
* Uncontrolled infection (i.e., progressive symptoms related to infection despite treatment or persistently positive microbiological cultures despite treatment or any other evidence of severe sepsis)
* Severe organ dysfunction within 3 days of enrollment including requirement for dialysis, mechanical ventilation, continuous BiPAP, or continuous high flow oxygen by nasal cannula, or total bilirubin ≥ 3x upper limit of normal not due to GVHD.
* A clinical presentation resembling de novo chronic GVHD or overlap syndrome developing before or present at the time of enrollment (except for mild oral or ocular GVHD)
* Corticosteroids >10 mg/day methylprednisolone (or other methylprednisolone equivalent, MPE) for any indication within 5 days before the onset of acute GVHD except for adrenal insufficiency or premedication for transfusions/IV meds
* Participation in clinical trials using experimental agents not approved by the FDA for any indication within 14 days of enrollment or five half-lives, whichever is longer provided any prior adverse events have improved to ≤grade 1
* Patients who are pregnant or nursing
* History of allergic reaction to ruxolitinib or any JAK inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-04-14 (Estimated)

PRIMARY OUTCOMES:
Day 28 Treatment Response | 28 days
  Day 28 response to treatment defined as complete (CR), very good partial (VGPR), or partial (PR) response without intervening therapy or death to ruxolitinib monotherapy.
  CR - All evaluable organs (skin, liver, GI tract) stage 0. For a response to be scored as CR, the patient must be in CR on the date of assessment and have had no intervening additional GVHD therapy.
  VGPR - Stage 0 liver and GI and residual stage 1 skin GVHD. For a response to be scored as VGPR, the patient must be in VGPR on the date of assessment and have had no intervening additional GVHD therapy.
  PR - An improvement by one or more stages in one or more organ involved with GVHD symptoms without worsening in others. For a response to be scored as PR, the patient must be in PR on the date of assessment and have had no intervening additional GVHD therapy.

SECONDARY OUTCOMES:
Steroid-refractory GVHD | 28 days
  Steroid Refractory (SR) GVHD is defined as GVHD that either does not achieve a clinical response or an additional line of therapy is initiated by day 28 from the initiation of systemic steroid therapy for non-responsive GVHD.
Durable response at day 56 | 56 days
  Durable response at day 56 is defined as CR, VGPR, or PR by day 28 and no GVHD flare, intervening treatment or death by day 56
GVHD flares | 90 days
  Flare is defined as an increase in acute GVHD severity in at least one target organ by at least one stage that is treated with an additional line of treatment or an increase in steroid dose in methylprednisolone equivalents (MPE) by at least 25%
Cumulative systemic corticosteroid dose | 90 days
Chronic GVHD requiring systemic steroid treatment | 1 year
Overall survival | 1 year
  OS (overall survival) - defined as the time from the enrollment to death
Non-relapse mortality | 1 year
  Non-relapse mortality (NRM) - defined as any death that occurs after HCT not attributable to relapse of the underlying disease for transplant
Relapse | 1 year
  Relapse - defined as reoccurrence of the underlying disease for transplant

CONTACTS AND LOCATIONS:
Overall Officials: John Levine, MD, MS, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (11):
- United States (11):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Ohio State University, Columbus, Ohio
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Patient did not consent to this